CLINICAL TRIAL: NCT01061593
Title: Phase III, Double-blind, Placebo-controlled, Randomized, 1-month Clinical Trial of Immunoxel Combined With Anti-TB Therapy Versus Anti-TB Therapy With Placebo
Brief Title: Adjunct Immunotherapy With Immunoxel in Patients With TB and TB/HIV
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Lisichansk Regional Tuberculosis Dispensary (Other)
Collaborators: Ekomed LLC (Industry)
Responsible Party: Principal Investigator, Galyna Kutsyna, PI, Ekomed LLC
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LRTBD-2259
Record Dates: First submitted 2010-02-02; First posted 2010-02-03 (Estimated); Last update posted 2015-05-20 (Estimated); Status verified 2015-05

CONDITIONS: Tuberculosis; HIV
Keywords: TB; MDR-TB; XDR-TB; TB/HIV
MeSH Terms: conditions — Tuberculosis; Tuberculosis, Multidrug-Resistant; Extensively Drug-Resistant Tuberculosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ATT+Immunoxel (Experimental): TB patients with DS-TB, MDR-TB, XDR-TB or TB-HIV on standard ATT + Immunoxel honey lozenge once per day day
  Interventions: Dietary Supplement: Immunoxel
- ATT+Placebo (Placebo Comparator): TB patients with DS-TB, MDR-TB, XDR-TB or TB-HIV on standard ATT + Placebo lozenge made of corn syrup once/day
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Immunoxel — 1 lozenge once per day
  Other Names: Immunoxel honey lozenges
  Arms: ATT+Immunoxel
Other: Placebo — 1 lozenge once per day
  Other Names: Placebo lozenge
  Arms: ATT+Placebo

SUMMARY:
Dzherelo (Immunoxel) is an oral immunomodulating botanical agent available over-the-counter in Ukraine. After many years of laboratory and clinical testing the formulation was approved in 1997 by the Ministry of Health of Ukraine as a dietary herbal supplement, which enhances immunity against viral and infectious diseases. The goal of this study is to conduct confirmatory clinical trial in Ukraine and Mongolia for TB indications.

DETAILED DESCRIPTION:
Phase III, placebo-controlled trial, aimed to seek the therapeutic benefit of Immunoxel in combination with standard of care anti-TB therapy (ATT) at the end of the 1-month period (p<0.05) among subjects with sputum-positive pulmonary TB. The results will be compared to standard ATT therapy + placebo. The trial will consist of one stage with laboratory evaluation after one month. Two cohorts or arms of at least 150 subjects each (total 300) with pulmonary TB positive for sputum AFB smear will be randomized in a 1:1 ratio to receive once-daily, honey lozenge of Immunoxel in combination with standard ATT for 1 month. Patients who receive standard ATT + placebo preparation will be used as a group of comparison.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are at least 18 years and are willing and capable of providing informed consent. Both men and non-pregnant women will be included. One group of at least 30 patients will have HIV. Another group of at least 30 patients will have MDR-TB. Another group of at least 30 patients will have XDR-TB Remaining patients will have drug-sensitive TB. They will be randomly assigned to placebo at 1:1 ratio.
* TB infection documented prior to Study Entry by sputum smear positive staining for acid-fast bacilli (AFB).
* Agreement to participate in the study and to give a sample of blood for HIV testing if required.
* Readily available home or other address where patient can be easily found at follow-up studies.

Exclusion Criteria:

* Subjects who have already taken Immunoxel in prior trials and those without sufficient baseline data. Those who met inclusion criteria can be retrospectively enrolled. Those who are re-treated and relapsed will be eligible as long as they are on the same drug regimen as the rest of patients. Pregnant or breast-feeding women are excluded.
* Subjects who have taken anti-retroviral drugs or immunomodulatory therapies within 2 months prior to Entry: systemic corticosteroids, immune globulin (IV gamma globulin, IVIG), interferons, interleukins, pentoxifylline (Trental), thalidomide, filgrastim (G-CSF), sargramostim (GM-CSF); dinitrochlorobenzene (DNCB), thymosin alpha 1 (thymosin alpha), thymopentin, inosiplex (Isoprinosine), polyribonucleoside (Ampligen), ditiocarb sodium (Imuthiol), any locally available immune modulators, and any other therapeutic or preventive vaccine. Subjects requiring concurrent participation in another experimental research treatment study, or who received an experimental agent within four weeks prior to Study Entry.
* History of angina, cardiac arrhythmias, clinically significant electrocardiogram abnormalities, or congestive heart failure. Evidence of active or acute cardiac disease, concomitant hypertension, epilepsy, or serious forms of extra-pulmonary tuberculosis.
* History of malignancy, other than minimal Kaposi sarcoma or other localized skin cancer (e.g. <10 cutaneous lesions, no evidence of visceral KS, etc.), or who have had prior cancer chemotherapy.
* Medical conditions that in the opinion of the local investigator, may obscure the proper observation of the safety or activity of the study treatment; including any acute medical condition of unknown etiology or recent surgery prior to Entry.
* Medical conditions such as active alcohol or substance abuse, or psychological issues that in the opinion of the local investigator, would interfere with adherence to the requirements of this study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 269 (Actual)
Dates: Start 2010-01; Primary Completion 2015-03 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
To compare the efficacy of combination of Immunoxel with anti-TB treatment versus anti-TB treatment with placebo in adults with sputum smear positive pulmonary tuberculosis | 1 month

SECONDARY OUTCOMES:
To confirm the safety of Immunoxel as demonstrated by Liver functions tests (ALT and bilirubin) and hemoglobin; effect on TB-associated wasting by measuring body weight. Effect on lymphocytes and CD4+ cells, CD4/CD8 ratio among those who have HIV. | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Galyna kutsyna, MD, PhD, Principal Investigator — Ekomed LLC
Locations (2):
- Misheel Lung surgery hospital,, Ulaanbaatar, Ulaanbaatar, Mongolia
- Kharkiv Medical National University, Kharkiv, Ukraine, Ukraine

REFERENCES:
- [Result] Efremenko YV, Arjanova OV, Prihoda ND, Yurchenko LV, Sokolenko NI, Mospan IV, Pylypchuk VS, Rowe J, Jirathitikal V, Bourinbaiar AS, Kutsyna GA. Clinical validation of sublingual formulations of Immunoxel (Dzherelo) as an adjuvant immunotherapy in treatment of TB patients. Immunotherapy. 2012 Mar;4(3):273-82. doi: 10.2217/imt.11.176. PMID 22401633
- [Result] Bourinbaiar AS, Mezentseva MV, Butov DA, Nyasulu PS, Efremenko YV, Jirathitikal V, Mishchenko VV, Kutsyna GA. Immune approaches in tuberculosis therapy: a brief overview. Expert Rev Anti Infect Ther. 2012 Mar;10(3):381-9. doi: 10.1586/eri.12.1. PMID 22397570
- [Derived] Batbold U, Butov DO, Kutsyna GA, Damdinpurev N, Grinishina EA, Mijiddorj O, Kovolev ME, Baasanjav K, Butova TS, Sandagdorj M, Batbold O, Tseveendorj A, Chunt E, Zaitzeva SI, Stepanenko HL, Makeeva NI, Mospan IV, Pylypchuk VS, Rowe JL, Nyasulu P, Jirathitikal V, Bain AI, Tarakanovskaya MG, Bourinbaiar AS. Double-blind, placebo-controlled, 1:1 randomized Phase III clinical trial of Immunoxel honey lozenges as an adjunct immunotherapy in 269 patients with pulmonary tuberculosis. Immunotherapy. 2017 Jan;9(1):13-24. doi: 10.2217/imt-2016-0079. Epub 2016 Nov 21. PMID 27868466
- See also: Enhancement of efficacy of tuberculosis drugs with Immunoxel (Dzherelo) in HIV-infected patients with active pulmonary tuberculosis. — http://www.ncbi.nlm.nih.gov/pubmed/20635986
- See also: Changes in CD4+ T-cells and HIV RNA resulting from combination of anti-TB therapy with Dzherelo in TB/HIV dually infected patients. — http://www.ncbi.nlm.nih.gov/pubmed/19920896
- See also: Effect of Immunomodulating Adjuvant Dzherelo (Immunoxel) in HIV Infected Patients Receiving Standard Antiretroviral Therapy. — http://www.ncbi.nlm.nih.gov/pubmed/19572055
- See also: Synthetic and natural immunomodulators acting as interferon inducers. — http://www.ncbi.nlm.nih.gov/pubmed/19355963
- See also: Cytokine profiles of HIV patients with pulmonary tuberculosis resulting from adjunct immunotherapy with herbal phytoconcentrates Dzherelo and Anemin. — http://www.ncbi.nlm.nih.gov/pubmed/19027322